CLINICAL TRIAL: NCT03908346
Title: A Novel Patient Decision Aid for Surrogate Decision Makers of Comatose Survivors of Cardiac Arrest: A Pilot Study
Brief Title: A Novel Patient Decision Aid for Surrogate Decision Makers of Comatose Survivors of Cardiac Arrest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Emergency Medicine Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-0795; K23HL138164 (NIH); EMF20_MCRD_00007 (Other Grant/Funding Number: Emergency Medicine Foundation)
Record Dates: First submitted 2019-04-04; First posted 2019-04-09 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Cardiac Arrest With Successful Resuscitation
Keywords: Neurologic Prognosis; Guideline Concordance; Surrogate Decision Makers
MeSH Terms: interventions — Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Decision Aid for Surrogate Decision Makers (Other): In this pilot trial all participants will be presented with the decision aid and queried as to the feasibility, acceptability and knowledge translation that is gained by exposure to the decision aid
  Interventions: Other: Decision Aid for Surrogate Decision Makers of Comatose Survivors of Cardiac Arrest

INTERVENTIONS:
Other: Decision Aid for Surrogate Decision Makers of Comatose Survivors of Cardiac Arrest — a decision aid has been created that is a four page document meant to support surrogate decision makers for comatose survivors of cardiac arrest

SUMMARY:
This study will test the feasibility and acceptability of deploying a decision aid for surrogate decision makers of comatose survivors of cardiac arrest early during hospitalization. This decision aid is to inform, educate and support decision makers charged with determining goals of care during post-cardiac arrest treatment.

DETAILED DESCRIPTION:
Survival and neurological recovery after out-of-hospital cardiac arrest are highly variable, driven in part by inconsistent hospital care following successful resuscitation. International guidelines for post-cardiac arrest care recommend delaying neurologic prognostication until 72-hours after resuscitation because early prognostication is imprecise and may precipitate inappropriate withdrawal of life sustaining therapy (WLST). Early WLST has been observed in-post cardiac arrest care. In order to encourage better guideline concordant care, the study proposes the implementation of an educational tool to support and inform surrogate decision makers in post-cardiac arrest care and neuro-prognostication. This pilot study will test the feasibility of implementing an educational tool for surrogate decision makers, the acceptability of such an intervention and early measures of knowledge translation. This study will inform the creation of a randomized controlled trial to test the ability of the tool to encourage guideline concordant timing of post-cardiac arrest neuro-prognostication.

ELIGIBILITY:
Inclusion Criteria:

* Adult 18 years of age and older
* Identified as a surrogate decision maker for patient who is a comatose survivor of out of hospital cardiac arrest

Exclusion Criteria:

* Illiterate or poor proficiency (unable to read decision aid)
* Non-english speaking

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2020-07-21 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Reach | Through study completion, on average 2.5 years
  To establish Reach, the investigators will determine the following: (1) number of out-of hospital cardiac arrests that present to the University of Colorado Hospital (UCH) ED; (2) number of Out of Hospital Cardiac Arrest (OHCA) patients with family/surrogate decision makers in the ED; (3) number of surrogate decision makers who agree to participate. Establishing reach is integral as it will allow us to determine the feasibility of intervening in the ED and will characterize the difficulties enrolling decision makers. The research assistant will keep a running tabulation of these data.
Effectiveness - Knowledge | Through study completion, on average 2.5 years
  Determine the number of individuals who reviewed the educational tool and completed the follow up knowledge evaluation. The pre-knowledge and post-knowledge/acceptability surveys will establish how effective the tool was at relaying information to the surrogate decision maker.
Adoption | Through study completion, on average 2.5 years
  To maximize adoption, 8-10 qualitative interviews will be conducted with emergency medicine providers, nurses and ancillary staff to explore barriers to use and potential adaptations to the implementation that might improve real world use. Providers who did not deploy the device will be included in order to understand their reasons for not adopting the intervention. Surrogate decision makers who did not agree to participate in the pilot intervention will be queried to understand their reasons for non-participation.
Implementation | Through study completion, on average 2.5 years
  In order to assess implementation (and prepare for larger implementation) a work-flow analysis will be conducted of the post-cardiac educational tools within the UCH ED. Nurses, ancillary staff (chaplain, social worker) who participate in family meetings within the emergency department will be queried. Via work-flow analysis, an understanding will be gained about when the tool was deployed, potential barriers/facilitators to deployment and how to best implement in a busy ED.

SECONDARY OUTCOMES:
Effectiveness - Patient Outcomes | Through study completion, on average 2.5 years
  As a secondary outcome, outcomes data for the cardiac arrest patients will be measured. These data will include the disposition, including withdrawal of life sustaining therapy, survival, or re-arrest.
Effectiveness - Decision Quality | Through study completion, on average 2.5 years
  We will measure decision regret using the Ottawa decision Regret Scale, decision conflict, emotional distress using promis measures and self efficacy using a validated scale derived for surrogate decision makers. This data will measure decision quality as a result of the tool.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States